CLINICAL TRIAL: NCT05171114
Title: Scleroderma: Description of Functional Disability Between the Dominant and Contralateral Hand, a Single-centre Descriptive Cohort.
Brief Title: Scleroderma: Functional Disability Between the Dominant and Contralateral Hand.
Acronym: SCLERO-HAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 87RI21_0029
Record Dates: First submitted 2021-11-29; First posted 2021-12-28 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Scleroderma, Systemic
Keywords: scleroderma; dermatology
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: Prospective, descriptive and comparative, monocentric pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate Scleroderma (Experimental): Patients with Cochin hand score less than or equal to 16
  Interventions: Diagnostic Test: Measurement of joint amplitudes
- severe Scleroderma (Experimental): Patients with Cochin hand score greater than 16
  Interventions: Diagnostic Test: Measurement of joint amplitudes

INTERVENTIONS:
Diagnostic Test: Measurement of joint amplitudes — Measurement of joint amplitudes by goniometry of the MCP, IPP, IPD for 2, 3, 4 and 5th radii, 1st commissure spacing and Kapandji score for the thumb

SUMMARY:
Systemic sclerosis is an autoimmune disease in which the hand is responsible for 75% of the overall disability. Management is based on systemic treatments combined with kinesitherapy aimed at maintaining joint amplitudes, improving muscle strength and preventing stiffness. The aim of this study is to describe and compare the average spontaneous and attempted reduction range of motion limitations between the dominant and contralateral hand.

DETAILED DESCRIPTION:
Systemic sclerosis is an autoimmune disease in which the hand is responsible for 75% of the overall disability. In case of limitation, the level of skin fibrosis, Raynaud's syndrome and its complications, the search for painful joints with or without synovitis, and the presence of calcifications must therefore be assessed. Management is based on systemic treatments combined with kinesitherapy aimed at maintaining joint amplitudes, improving muscle strength and preventing stiffness. No study to date has compared the functionality of one hand to the other. The hypothesis is that there is a difference in range of motion limitations between the dominant hand and the contralateral hand.

Patients in the active file of the Internal Medicine A department of the Limoges University Hospital who meet the inclusion criteria will be offered the study by telephone. Patients wishing to participate will be given an appointment on a dedicated consultation slot. During this visit, Patients will be given an information note and their consent will be collected. The study examinations will be performed and the questionnaire completed. At the end of this visit, the study will be completed for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 :
* Major patient
* Diagnosis of diffuse or limited cutaneous systemic sclerosis according to the new ACR/EULAR criteria
* Cochin hand score less than or equal to 16
* Group 2 :
* Major patient
* Diagnosis of diffuse or limited cutaneous systemic sclerosis according to the new ACR/EULAR criteria
* Cochin hand score greater than 16.

Exclusion Criteria:

* Overlap syndrome (Sharp or scleromyositis 2)
* Patient with another autoimmune disease
* History of surgery or trauma to the hand with proven functional sequelae
* Presence of synovitis
* Patient with Dupuytren's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Measurement of joint amplitudes | at inclusion
  Measurement of joint amplitudes by goniometry

SECONDARY OUTCOMES:
Digital skin score | at inclusion
  Measure with modified Rodnan skin score. The value of this score varies from 0 (no cuntaneous sclerosis) to 51(severe cutaneous sclerosis).
Digital pressure | at inclusion
  use of Finger Systolic Blood Pressure Index (FBPI) proposed by Blaise et al.
Number of digital ulcers | at inclusion
Number of subcutaneous calcifications | at inclusion
Visual Analog Score for pain | at inclusion
  Score varie from 0 (no pain) to 10 (worst pain possible)
number of painful joints | at inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France